CLINICAL TRIAL: NCT02663544
Title: The Impact of Low-fat and Full-fat Dairy Consumption on Glucose Homeostasis (DAIRY Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Mario Kratz, Associate Member, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DRI2395
Record Dates: First submitted 2016-01-21; First posted 2016-01-26 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Insulin Resistance; Metabolic Syndrome; Obesity; Diabetes; NAFLD; Inflammation
Keywords: Diabetes; Metabolic syndrome; Obesity; NAFLD
MeSH Terms: conditions — Insulin Resistance; Metabolic Syndrome; Obesity; Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Limited dairy diet (Active Comparator): Three 8 oz. servings per week of non-fat milk. Participants will otherwise eat their usual diet, but will be asked not to consume any dairy products not provided by the study.
  Interventions: Other: Limited dairy diet
- Low-fat dairy diet (Experimental): 3.3 daily servings of non-fat and low-fat dairy products in the form of fluid milk, cheese and yogurt. Participants will otherwise eat their usual diet, and will be asked not to consume any dairy products not provided by the study.
  Interventions: Other: Low-fat dairy diet
- Full-fat dairy diet (Experimental): 3.3 daily servings of full-fat dairy products in the form of fluid milk, cheese and yogurt. Participants will otherwise eat their usual diet, and will be asked not to consume any dairy products not provided by the study.
  Interventions: Other: Full-fat dairy diet

INTERVENTIONS:
Other: Limited dairy diet — Consumption of no dairy foods other than 3 servings per week of nonfat milk for 12 weeks
  Arms: Limited dairy diet
Other: Low-fat dairy diet — Consumption of 3.3 servings per day of low-fat milk, yogurt, and cheese for 12 weeks
  Arms: Low-fat dairy diet
Other: Full-fat dairy diet — Consumption of 3.3 servings per day of full-fat milk, yogurt, and cheese for 12 weeks
  Arms: Full-fat dairy diet

SUMMARY:
This randomized controlled feeding trial aims to determine whether the consumption of different amounts and types of dairy products affects blood sugar regulation and cardiometabolic health in men and women with the metabolic syndrome.

DETAILED DESCRIPTION:
This is a randomized controlled feeding trial designed to investigate whether the consumption of a diet rich in low-fat dairy vs. full-fat dairy vs. a limited dairy diet differentially affects glucose homeostasis. The researchers will also begin an investigation into the mechanisms by which dairy may affect glucose tolerance and its determinants. The investigators will study 60 men and women with the metabolic syndrome who will consume diets differing in their type and content of dairy foods, in a parallel-design randomized controlled trial consisting of a 4-week wash-in diet period and a 12-week dietary intervention period.

Subjects will be randomized using block randomization stratified by gender and insulin resistance (low insulin resistance vs. high insulin resistance or manifest diabetes) to one of three diet groups, which they will follow for 12 weeks: the limited dairy diet, the low-fat dairy diet, or the full-fat dairy diet. During the dietary intervention, participants will be provided with specific amounts and types of dairy products by the Human Nutrition Lab (HNL) at Fred Hutchinson Cancer Research Center (FHCRC). In the limited dairy diet arm, participants will be asked not to consume any dairy, other than three servings of nonfat milk per week, which will be provided. In the two dairy diet arms, participants will be asked to consume 3.3 servings per day of either nonfat/low-fat or full-fat milk, yogurt, and cheese. Participants will be asked to consume all of the dairy products they receive, not to consume any other dairy products for 12 weeks, and to continue consuming their habitual diet ad libitum (i.e., to eat only when hungry, and to stop eating when comfortably satiated).

Prior to randomization, subjects will complete a wash-in diet period of 4 weeks during which they will be asked to consume the limited dairy diet (i.e., consume 3 servings of nonfat milk per week, and not consume any other dairy products). In the third week of the wash-in diet period, subjects will also complete their first of two 5-day controlled feeding periods (i.e., consume study dairy products alongside a provided standard American diet) to measure ad libitum energy intake. During the last week of the wash-in diet period, participants will be admitted to clinic for a baseline visit (clinic visit #1). After clinic visit #1, subjects will be randomized to one of the three study arms, as outlined above. They will follow their randomly assigned study diet for the next 12 weeks. In the second week of the main intervention period, subjects will complete their second 5-day controlled feeding period to again measure ad libitum energy intake, this time on the specific intervention diet they had been randomized to. In the last week of the 12-week diet phase, subjects will be admitted for the follow-up clinic visit (clinic visit #2). At both clinic visits, the researchers will collect fasting blood; measure body weight and height, waist and hip circumference, and blood pressure; conduct a 3-hour FS-OGTT to assess glucose tolerance, insulin sensitivity, and pancreatic beta-cell function; conduct a whole-body DEXA scan to assess body fat mass, lean mass, and body fat distribution; and an abdominal MRI scan to assess liver triglyceride content and the ratio of intra-abdominal to subcutaneous adipose tissue. Subjects will also complete five Food Frequency Questionnaires (FFQ's) and five unannounced 24-hour dietary recalls during the study to assess dietary intakes.

The primary analysis will be a per protocol analysis that will include at least 60 participants (at least 20 in each intervention arm) who comply with all study procedures per protocol. The investigators anticipate enrolling up to 72 participants to achieve this goal. In a secondary analysis, the researchers will analyze the impact of the dietary intervention on all enrolled participants, including those who dropped out, were excluded, or non-compliant with the study protocol, in an intent-to-treat (ITT) analysis that will be reported and interpreted together with the per protocol analysis.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic syndrome (three of the following five criteria):

  * Increased waist circumference: In Asians: ≥ 90 cm in men, ≥ 80 cm in women; in all other races: ≥ 102 cm in men, ≥ 88 cm in women
  * Fasting plasma triglycerides ≥ 150 mg/dL, or drug treatment for elevated triglycerides
  * High-density lipoprotein (HDL)-cholesterol <40 mg/dL in males or <50 mg/dL in females, or drug treatment for reduced HDL-cholesterol
  * Systolic blood pressure ≥ 135 mm Hg or diastolic blood pressure ≥ 85 mm Hg or drug treatment for hypertension
  * Fasting plasma glucose ≥ 100 mg/dL or previous diagnosis of diabetes
* Body weight within 10% of current weight over the last 6 months before starting the study
* Able to come to the FHCRC regularly to pick up food
* Able and willing to attend a study initiation meeting of ~1.5 hour duration at the FHCRC, two clinic visits of ~5 hours duration each at the University of Washington (UW) Medial Center Clinical Research Center (CRC), and two clinic visits of ~2 hours duration each at the UW Bio-Molecular Imaging Center (BMIC)
* Willing to follow the dietary regimen
* Able to provide informed consent

Exclusion Criteria:

* Antidiabetic medications or insulin within the last 6 months
* Uncontrolled diabetes, defined as HbA1c > 8.0%
* Allergy to milk protein
* Presence of major chronic inflammatory or autoimmune disease (with acute symptoms or CRP > 10 mg/L), or malabsorption syndromes
* Presence or history of liver disease or end-stage renal disease requiring dialysis
* Uncontrolled thyroid disease
* Inability or unwillingness to eat the provided foods
* Contraindications for MRI scan other than body size
* Intake of drugs likely to interfere with study endpoints, including corticosteroids, anabolic steroids, antiretroviral drugs, anti-psychotic drugs and immunosuppressive drugs (within 3 months of starting the study)
* Regular high-dose use of non-steroidal anti-inflammatory drugs (more than 3 times per week and more than 600 mg per day, within 3 months of starting the study)
* Presence or recent history of anemia (within 3 months of starting the study)
* History of bariatric surgery
* Participation in an intervention study or weight-loss program (within 3 months of starting the study)
* Alcohol intake > 2 drinks per day (within 12 months of starting the study)
* Use of tobacco products, eCigarettes, or recreational drugs on more than 2 days per month (within 12 months of starting the study)
* Current or recent (within 12 months of starting the study) pregnancy or breastfeeding, or intention of becoming pregnant in the next 6 months
* Fasting Triglycerides >1000mg/dL
* Any cancer other than non-melanoma skin cancer in the last 3 years
* Other significant health condition, as determined by researcher and Physician of Record, that makes the individual unfit to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01; Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Change in glucose tolerance | Difference between pre- and post 12-week intervention period
  As measured by glucose area under the curve during a frequently sampled 3-hour oral glucose tolerance test (FS-OGTT).

SECONDARY OUTCOMES:
Change in systemic insulin sensitivity | Difference between pre- and post 12-week intervention period
  As measured by the Matsuda-De Fronzo Insulin Sensitivity Index based on the FS-OGTT
Change in pancreatic beta-cell function: insulinogenic index | Difference between pre- and post 12-week intervention period
  As measured by the insulinogenic index based on the FS-OGTT
Change in pancreatic beta-cell function: oral disposition index | Difference between pre- and post 12-week intervention period
  As measured by the oral disposition index (DI), the product of insulin sensitivity (Matsuda-De Fronzo index) and beta-cell function (insulinogenic index)
Change in liver fat content | Difference between pre- and post 12-week intervention period
  As measured by an abdominal magnetic resonance imaging (MRI) scan
Change in low-grade chronic systemic inflammation: hsCRP | Difference between pre- and post 12-week intervention period
  As measured by fasting plasma concentration of C-reactive protein (CRP)
Change in low-grade chronic systemic inflammation: IL-6 | Difference between pre- and post 12-week intervention period
  As measured by fasting plasma concentration of interleukin-6 (IL-6)
Change in pancreatic beta-cell function: glucose sensitivity | Difference between pre- and post 12-week intervention period
  Glucose sensitivity, as modeled from the glucose, insulin, and c-peptide data obtained from the FS-OGTT

OTHER OUTCOMES:
Change in total body fat mass | Difference between pre- and post 12-week intervention period
  Total body fat mass (kg), as measured by whole body dual-energy x-ray absorptiometry (DEXA) scan
Change in abdominal fat mass | Difference between pre- and post 12-week intervention period
  Abdominal fat mass (kg), as measured by whole body dual-energy x-ray absorptiometry (DEXA) scan
Change in abdominal subcutaneous-to-visceral fat ratio | Difference between pre- and post 12-week intervention period
  Abdominal subcutaneous-to-visceral fat ratio, as measured by abdominal magnetic resonance imaging (MRI) scan
Change in body weight | Difference between pre- and post 12-week intervention period
  Body weight will be measured on a calibrated digital scale in kilogram (kg) while wearing a hospital gown
Change in average diurnal glucose concentrations | Difference between pre- and post 12-week intervention period
  The average diurnal glucose concentration will be assessed by measuring hemoglobin A1c (HbA1c)
Change in fasting glucose concentration | Difference between pre- and post 12-week intervention period
  Glucose concentration (mg/dL) will be measured in fasting plasma
Change in systolic blood pressure | Difference between pre- and post 12-week intervention period
  Systolic blood pressure (mmHg), as measured following the American Heart Association blood pressure protocol
Change in diastolic blood pressure | Difference between pre- and post 12-week intervention period
  Diastolic blood pressure (mmHg), as measured following the American Heart Association blood pressure protocol
Change in ad libitum energy intake over 5 days | Difference in energy intake during a 5-day controlled feeding period in the study wash-in period as compared to a 5-day controlled feeding period in the intervention period
  Ad libitum energy intake will be assessed during two 5-day ad libitum controlled feeding periods
Change in fasting serum total cholesterol concentration | Difference between pre- and post 12-week intervention period
  The total cholesterol concentration (mg/dL) will be measured in fasting serum
Change in fasting serum high-density lipoprotein (HDL) cholesterol concentration | Difference between pre- and post 12-week intervention period
  The cholesterol concentration in HDL (mg/dL) will be measured in fasting serum
Change in fasting serum triglyceride concentration | Difference between pre- and post 12-week intervention period
  The triglyceride concentration (mg/dL) will be measured in fasting serum
Change in fasting serum low-density lipoprotein (LDL) cholesterol concentration | Difference between pre- and post 12-week intervention period
  The cholesterol concentration in LDL (mg/dL) will be measured in fasting serum, or calculated by the Friedewald formula
Change in cholesterol concentration in 38 serum lipoprotein fractions | Difference between pre- and post 12-week intervention period
  As assessed by measuring the cholesterol content (mg/dL) in 38 lipoprotein fractions isolated from fasting serum by KBr gradient ultracentrifugation
Change in fasting plasma total adiponectin | Difference between pre- and post 12-week intervention period
  The total adiponectin concentration (ug/mL) will be measured in fasting plasma
Change in waist circumference | Difference between pre- and post 12-week intervention period
  Waist circumference (cm)
Change in hip circumference | Difference between pre- and post 12-week intervention period
  Hip circumference (cm)
Change in the waist-to-hip-ratio | Difference between pre- and post 12-week intervention period
  Ratio of waist circumference (cm) to hip circumference (cm)
Change in trunk fat mass | Difference between pre- and post 12-week intervention period
  Trunk fat mass (kg), as measured by dual-energy x-ray absorptiometry (DEXA)-scan
Change in peripheral fat mass | Difference between pre- and post 12-week intervention period
  Peripheral fat mass (kg), defined as the fat mass of all limbs, as measured by dual-energy x-ray absorptiometry (DEXA)-scan
Change in visceral fat mass | Difference between pre- and post 12-week intervention period
  Visceral fat mass (inches^2), as estimated by dual-energy x-ray absorptiometry (DEXA)-scan
Change in the low-density lipoprotein (LDL) relative flotation rate | Difference between pre- and post 12-week intervention period
  The LDL relative flotation rate (Rf) is calculated as the fraction number of the major peak of LDL divided by the total number of fractions
Change in fasting insulin concentration | Difference between pre- and post 12-week intervention period
  The insulin concentration (uU/L) measured in fasting plasma
Change in the homeostasis model assessment (HOMA) insulin resistance index | Difference between pre- and post 12-week intervention period
  The HOMA insulin resistance index will be calculated from glucose and insulin concentrations measured in fasting plasma

CONTACTS AND LOCATIONS:
Overall Officials: Mario Kratz, PhD, Principal Investigator — Fred Hutchinson Cancer Research Center, Associate Member
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized blood samples and study data may be shared with outside investigators who sign confidentiality pledges (from participants who have given written consent for the use of study specimen and data for 'other research' only).

REFERENCES:
- [Derived] Fernando I, Schmidt KA, Cromer G, Burhans MS, Kuzma JN, Hagman DK, Utzschneider KM, Holte S, Kraft J, Vaughan TL, Kratz M. The impact of low-fat and full-fat dairy foods on symptoms of gastroesophageal reflux disease: an exploratory analysis based on a randomized controlled trial. Eur J Nutr. 2022 Aug;61(5):2815-2823. doi: 10.1007/s00394-022-02855-6. Epub 2022 Mar 16. PMID 35294608
- [Derived] Schmidt KA, Cromer G, Burhans MS, Kuzma JN, Hagman DK, Fernando I, Murray M, Utzschneider KM, Holte S, Kraft J, Kratz M. Impact of low-fat and full-fat dairy foods on fasting lipid profile and blood pressure: exploratory endpoints of a randomized controlled trial. Am J Clin Nutr. 2021 Sep 1;114(3):882-892. doi: 10.1093/ajcn/nqab131. PMID 34258627
- [Derived] Schmidt KA, Cromer G, Burhans MS, Kuzma JN, Hagman DK, Fernando I, Murray M, Utzschneider KM, Holte S, Kraft J, Kratz M. The impact of diets rich in low-fat or full-fat dairy on glucose tolerance and its determinants: a randomized controlled trial. Am J Clin Nutr. 2021 Mar 11;113(3):534-547. doi: 10.1093/ajcn/nqaa301. PMID 33184632